CLINICAL TRIAL: NCT04176588
Title: A Phase 3, Randomized, Placebo-Controlled, Double-Blind, Multicenter Study to Evaluate the Efficacy and Safety of Etrasimod for Induction and Maintenance Treatment in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Phase 3 Study of Etrasimod in Subjects With Moderately to Severely Active Ulcerative Colitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Everstar Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ES101002
Record Dates: First submitted 2019-11-22; First posted 2019-11-25 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Moderately to Severely Active Ulcerative Colitis
MeSH Terms: interventions — etrasimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Etrasimod 2mg (Experimental): 2mg/tablet, administratered orally, once daily
  Interventions: Drug: Etrasimod
- Placebo Comparator: Placebo (Placebo Comparator): matching tablet, administratered orally, once daily
  Interventions: Drug: Placebo
- Etrasimod 2mg (optional open-label extension period) (Experimental): 2mg/tablet, administratered orally, once daily
  Interventions: Drug: Etrasimod

INTERVENTIONS:
Drug: Etrasimod — Drug:Etrasimod Tablet other name:APD334
  Arms: Etrasimod 2mg (optional open-label extension period); Experimental: Etrasimod 2mg
Drug: Placebo — Drug:placebo Tablet
  Arms: Placebo Comparator: Placebo

SUMMARY:
The purpose of this study is to determine whether etrasimod is a safe and effective treatment for moderately to severely active ulcerative colitis.

Condition or disease: Ulcerative Colitis Intervention/treatment: Drug: Etrasimod Drug: Placebo Phase: Phase 3

ELIGIBILITY:
Inclusion Criteria:

1. A documented of diagnosis with UC at least 3 months prior to screening.
2. Have active UC confirmed by endoscopy with ≥ 10 cm rectal involved.

Exclusion Criteria:

1. Have severe extensive colitis
2. Diagnosis of Crohn's disease or indeterminate colitis or the presence or history of a fistula consistent with Crohn's disease
3. Diagnosis of microscopic colitis, ischemic colitis, infection colitis or colonic mucosal dysplasia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of Subjects With Clinical Remission Assessed by modified Mayo score(mMS) | induction period week 12
  Clinical remission per mMS(endoscopy, rectal bleeding, stool frequency), ranging from 0-9 (normal to severe)
Proportion of Subjects With Clinical Remission Assessed by modified Mayo score(mMS) | Maintenance period week 40
  Clinical remission per mMS, ranging from 0-9 (normal to severe)

SECONDARY OUTCOMES:
Proportion of Subjects Achieving Endoscopic Improvement Assessed by endoscopic subscore | induction period week 12
  Endoscopic improvement per endoscopy subscore, ranging from 0 to 3 (normal to severe)
Proportion of Subjects with Clinical Response Assessed by modified Mayo score(mMS) | induction period Week 12
  Clinical response per mMS, ranging from 0 to 9 (normal to severe).
Proportion of Subjects Achieving Endoscopic Improvement Assessed by endoscopic subscore | Maintenance period Week 40
  Endoscopic improvement per endoscopy subscore, ranging from 0 to 3 (normal to severe)
Proportion of Subjects with Clinical Response Assessed by modified Mayo score(mMS) | Maintenance period Week 40
  Clinical response per mMS, ranging from 0 to 9 (normal to severe)
Proportion of Subjects who achieve symptomatic response over time | Open label treatment period up to 40 Weeks
  Symptomatic response per paritial Mayo score(rectal bleeding, stool frequency), ranging from 0-6(normal to severe)
Proportion of Subjects who achieve Symptomatic Remission over time | Open label treatment period up to 40 Weeks
  Symptomatic remission per paritial Mayo score, ranging from 0-6(normal to severe)

CONTACTS AND LOCATIONS:
Overall Officials: Kaichun Wu, Principal Investigator — The First Affiliated Hospital of Fourth Military Medical University, PLA
Locations (1):
- The First Affiliated Hospital of Fourth Military Medical University, PLA, Xi’an, Shanxi, China

REFERENCES:
- [Derived] Wu K, Zheng C, Cao Q, Ding Y, Gao X, Zhong J, Chiu CT, Zhang H, Wang X, Wang B, Liang J, Liu X, Zhou Y, Xu B, Kim TO, Shen X, Chen D, Chen W, Liu Y, Shen J, Liu F, Ding X, Zhan Q, Chou JW, Zeng S, Lin Y, Ying L, Chen X; ENLIGHT UC Study Group. Etrasimod as induction and maintenance treatment for patients with moderately to severely active ulcerative colitis in East Asia (ENLIGHT UC): a randomised, double-blind, placebo-controlled, multicentre, phase 3 study. Lancet Gastroenterol Hepatol. 2025 Dec;10(12):1089-1103. doi: 10.1016/S2468-1253(25)00198-0. Epub 2025 Sep 30. PMID 41043449
- [Derived] Vermeire S, Rubin DT, Peyrin-Biroulet L, Dubinsky MC, Regueiro M, Irving PM, Goetsch M, Lazin K, Gu G, Wu J, Modesto I, McDonnell A, Guo X, Green J, Dalam AB, Yarur AJ. Cardiovascular events observed among patients in the etrasimod clinical programme: an integrated safety analysis of patients with moderately to severely active ulcerative colitis. BMJ Open Gastroenterol. 2025 Jan 8;12(1):e001516. doi: 10.1136/bmjgast-2024-001516. PMID 39778975